CLINICAL TRIAL: NCT06561698
Title: High-dose Dual Therapy and Minocycline-cotaining Quadruple Therapy for Helicobacter Pylori Infection
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hong Lu, MD, Medical Doctor of Division of Gastroenterology and Hepatology of Renji Hospital,Professor of Medicine, RenJi Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rjhy20240814
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-08

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; minocycline; amoxicillin
MeSH Terms: conditions — cyclopia sequence | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin; Minocycline; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dual therapy (Experimental)
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin
- Minocycline bismush quadruple therapy (Experimental)
  Interventions: Drug: Vonoprazan; Drug: Bismuth Potassium Citrate; Drug: Minocycline,Metronidazole

INTERVENTIONS:
Drug: Vonoprazan — Potassium competitive acid blocker
Drug: Amoxicillin — Antibiotics for H. pylori eradication
  Arms: Dual therapy
Drug: Bismuth Potassium Citrate — Gastric mucosal protective drug with anti-H. pylori effect
  Arms: Minocycline bismush quadruple therapy
Drug: Minocycline,Metronidazole — Antibiotics for H. pylori eradication
  Arms: Minocycline bismush quadruple therapy

SUMMARY:
This study is a multicentra, prospective study. The enrolled patients are HP positive. They are diagnosed as HP positive by rapid urease test and/or 13C urea breath test. According to the declaration of Helsinki, 200 patients will be included in this study. After obtaining the written informed consent of the patients, HP culture and drug sensitivity test will be conducted on all the selected patients with the success rate, adverse reactions, compliance, antibiotic resistance of HP and its impact on HP eradication.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to participate in the study and to sign and give informed consent
* Confirmed H. pylori infection

Exclusion Criteria:

* Pregnant and lactating women;
* History of gastrointestinal malignancies;
* History of previous subtotal gastrectomy;
* Serious dysfunction of heart, liver, kidney, lung and other important organs and congenital diseases; Such as grade IV cardiac insufficiency, liver failure, uremia, respiratory failure, hemophilia, Wilson disease, etc;
* History of hematological diseases
* People who are allergic to drugs;
* The guardian or patient refused to join the group;
* Alcohol and / or drug abuse (addiction or dependence) or poor compliance judged by doctors;
* No legal capacity or poor self-knowledge
* administration of antibiotics, bismuth, antisecretory drugs, or Chinese herb medicine in the preceding 8 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | Six weeks after completion of therapy
  Six weeks after completion of therapy, H. pylori eradication was assessed by ¹³C-urea breath test. Eradication was defined as negative result from urea breath test (<4‰) (4‰ as the cutoff value).

SECONDARY OUTCOMES:
Rate of adverse effects | Within 7 days after completion of therapy
  The subjects were asked to grade the severity of adverse events according to their influence on daily activities, experienced as "mild" (transient and well tolerated), "moderate" (causing discomfort and partially interfering with daily activities), or "severe" (causing considerable interference with daily activities)
Compliance rate | Within 7 days after completion of therapy
  Compliance was defined as poor when they had taken less than 80% of the total medication

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Hebi People's Hospital, Hebi, Henan
  - Jiaozuo People's Hospital, Jiaozuo, Henan
  - Luoyang central Hospital, Luoyang, Henan
  - The first people's hospital of ping ding shan, Pingdingshan, Henan
  - Xuchang central Hospital, Xuchang, Henan
  - The Second Affiliated Hospital of Henan University of science and technology, Zhengzhou, Henan
  - The Third People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Zhengzhou People's Hospital, Zhengzhou, Henan
  - Zhoukou Central Hospital, Zhoukou, Henan
  - Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality